CLINICAL TRIAL: NCT04270266
Title: Mind-Body Medicine for Adolescents and Young Adults (AYA) Coping With Lymphoma
Brief Title: Mind-Body Medicine for the Improvement of Quality of Life in Adolescents and Young Adults Coping With Lymphoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0282; NCI-2019-05846 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0282 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-09-12; First posted 2020-02-17 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Lymphoma
Keywords: All types of lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Early Intervention, Educational; Educational Status; Methods; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (meditation) (Experimental): Patients attend meditation group sessions over 75 minutes once weekly for up to 5 weeks.
  Interventions: Other: Meditation Therapy; Other: Questionnaire Administration
- Group II (educational) (Active Comparator): Patients attend educational group sessions over 75 minutes once weekly for up to 5 weeks.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Attend educational sessions
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group II (educational)
Other: Meditation Therapy — Attend meditation sessions
  Other Names: Meditation
  Arms: Group I (meditation)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well a mind-body intervention works in improving overall quality of life in adolescents and young adults with lymphoma. A meditation based mind-body intervention may help lower distress, depressive symptoms, and anxiety in adolescents and young adults coping with lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Examine the feasibility of the mind-body intervention in adolescents and young adults (AYAs) with lymphoma.

SECONDARY OBJECTIVE:

I. Establish the initial intervention efficacy regarding psychological distress and cancer symptoms (tertiary objective) relative to an attention control (AC) group.

EXPLORATORY OBJECTIVE:

I. Explore mediation (e.g., mindfulness, compassion, social connection, inflammatory processes) and moderation (e.g., demographic and medical factors) of the intervention effects.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients attend meditation group sessions over 75 minutes once weekly for up to 5 weeks.

GROUP II: Patients attend educational group sessions over 75 minutes once weekly for up to 5 weeks.

After completion of study intervention, patients are followed at 6 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 18-39 diagnosed within 6 months with stage I-IV Lymphoma (all types)
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or below
* Having access to the internet
* Able to read, write and speak English

Exclusion Criteria:

* Major psychiatric or cognitive deficits that would impede the completion of self-report instruments as deemed by the clinical team
* Regular (self-defined) participation in psychotherapy or a formal cancer support group

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2026-12-21 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Mind-body intervention in (AYAs) Adolescents and Young Adults with Lymphoma Questionnaire | Up to 12 weeks
  We will examine preliminary evidence of intervention efficacy. Meaning and Purpose (1-5) Strongly Disagree 1- Disagree 2, Neither agree or disagree 3, Agree 4, Strongly agree 5.
  Day-to-Day Experiences (1-6) Almost Always-1, Very frequently-2, Somewhat Frequently -3, Somewhat Infrequently-4, Very Infrequently-5, Almost Never 6

SECONDARY OUTCOMES:
Psychological distress and cancer symptoms (tertiary objective) relative to an attention control (AC) group Questionnaire | Up to 12 weeks
  We will examine preliminary evidence of intervention efficacy. Meaning and Purpose (1-5) Strongly Disagree 1- Disagree 2, Neither agree or disagree 3, Agree 4, Strongly agree 5.
  Day-to-Day Experiences (1-6) Almost Always-1, Very frequently-2, Somewhat Frequently -3, Somewhat Infrequently-4, Very Infrequently-5, Almost Never 6

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Cho D, Ahmed S, Snyder S, Kroll J, Chen M, Roth M, Milbury K. Group-Based Support Interventions for Adolescents and Young Adults With Lymphoma: A Pilot Randomized Controlled Trial. Psychooncology. 2025 Dec;34(12):e70343. doi: 10.1002/pon.70343. PMID 41298073
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org